CLINICAL TRIAL: NCT00042471
Title: Evaluation of the Bioavailability of Pramlintide
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 137-153
Record Dates: First submitted 2002-07-30; First posted 2002-08-01 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-08

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — pramlintide

ARMS (1):
- Pramlintide acetate (AC137) injection (Experimental): Pramlintide acetate (AC137) injection is a clear, colorless, sterile solution for injection. It consists of pramlintide in sodium acetate buffer, pH 4.0, containing 43mg/mL mannitol as an iso-osmolality modifier and 2.25 mg/mL metacresol as a preservative. The strength of pramlintide is 1.0 mg/mL for SC injection and 0.6 mg/mL for IV bolus injection.
  Interventions: Drug: Pramlintide acetate

INTERVENTIONS:
Drug: Pramlintide acetate — Pramlintide acetate (AC137) injection is a clear, colorless, sterile solution for injection. It consists of pramlintide in sodium acetate buffer, pH 4.0, containing 43mg/mL mannitol as an iso-osmolality modifier and 2.25 mg/mL metacresol as a preservative. The strength of pramlintide is 1.0 mg/mL for SC injection and 0.6 mg/mL for IV bolus injection.
  Other Names: Symlin (pramlintide acetate)

SUMMARY:
This is a randomized, open-label, crossover study to examine the bioavailability of pramlintide in normal weight and overweight subjects with type 1 and type 2 diabetes mellitus using insulin.

ELIGIBILITY:
Inclusion Criteria:

* HbA1c value between 6-12%
* BMI <= 27 kg/m2 or BMI >=30 to <= 45 kg/m2
* Consistent insulin regimen for 2 months prior to screening

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2002-06; Primary Completion 2002-12 (Actual); Study Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
Effect of varying needle length on bioavailability of Pramlintide | approximately 6days but not to exceed 14days
  To determine the effect of various anatomical injection sites and varying needle lengths upon the absolute bioavailability of pramlintide when injected subcutaneously (SC) in non-obese and obese subjects with type 1 and type 2 diabetes mellitus using insulin.

SECONDARY OUTCOMES:
Effect of varying needle length on safety and tolerability of Pramlintide | Approximately 6 days not to exceed 14days
  To assess the safety and tolerability of pramlintide when injected SC at various anatomical sites and with various needle lengths in non-obese and obese subjects with type 1 and type 2 diabetes mellitus using insulin

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Orlando Clinical Research Center, Orlando, Florida
  - New Orleans Center for Clinical Research, New Orleans, Louisiana
  - DaVita Clinical Research, Minneapolis, Minnesota
  - CEDRA Clinical Research, LLC, Austin, Texas